CLINICAL TRIAL: NCT03821402
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Dose-Ranging, Multi-Center Trial to Evaluate the Efficacy and Safety of DaxibotulinumtoxinA for Injection for the Treatment of Upper Limb Spasticity in Adults After Stroke or Traumatic Brain Injury
Brief Title: Efficacy and Safety of DaxibotulinumtoxinA for Injection for the Treatment of Adult Upper Limb Spasticity
Acronym: JUNIPER
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Revance Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1820203
Record Dates: First submitted 2019-01-15; First posted 2019-01-29 (Actual); Results first posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-08

CONDITIONS: Upper Limb Spasticity
Keywords: ULS; JUNIPER; DAXI for injection; Botulinum toxin
MeSH Terms: interventions — Injections

STUDY DESIGN:
Intervention Model Description: Eligible subjects will be randomized (1:1:1:1) to one of four treatment groups: Group 1: DAXI 250 U (N=32); Group 2: DAXI 375 U (N=32); Group 3: DAXI 500 U (N=32); Group 4: Placebo (N=32).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blinded. The subject, Sponsor, and study site research personnel will be blinded to the identity of the subject's assigned treatment.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- DAXI 250 U (Experimental): DAXI for injection for the treatment of Upper Limb Spasticity (ULS) in Adults with 250 U dose
  Interventions: Biological: DAXI for injection 250 U
- DAXI 375 U (Experimental): DAXI for injection for the treatment of Upper Limb Spasticity (ULS) in Adults with 375 U
  Interventions: Biological: DAXI for injection 375 U
- DAXI 500 U (Experimental): DAXI for injection for the treatment of Upper Limb Spasticity (ULS) in Adults with 500 U
  Interventions: Biological: DAXI for injection 500 U
- Placebo (Placebo Comparator): Placebo group
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: DAXI for injection 250 U — DaxibotulinumtoxinA for injection is a sterile, white to off-white lyophilized product containing the active ingredient, daxibotulinumtoxinA, and inactive ingredients to be reconstituted with sterile, non-preserved, 0.9% sodium chloride solution saline
  Arms: DAXI 250 U
Biological: DAXI for injection 375 U — DaxibotulinumtoxinA for injection is a sterile, white to off-white lyophilized product containing the active ingredient, daxibotulinumtoxinA, and inactive ingredients to be reconstituted with sterile, non-preserved, 0.9% sodium chloride solution saline.
  Arms: DAXI 375 U
Biological: DAXI for injection 500 U — DaxibotulinumtoxinA for injection is a sterile, white to off-white lyophilized product containing the active ingredient, daxibotulinumtoxinA, and inactive ingredients to be reconstituted with sterile, non-preserved, 0.9% sodium chloride solution saline
  Arms: DAXI 500 U
Other: Placebo — Placebo is a sterile lyophilized product consisting of inactive ingredients without the neurotoxin to be reconstituted with sterile, non-preserved 0.9% sodium chloride solution.
  Arms: Placebo

SUMMARY:
This is a randomized, Double-Blind, Placebo-Controlled, Parallel Group, Dose-Ranging, trial to Evaluate the Efficacy and Safety of DaxibotulinumtoxinA for Injection for the Treatment of Upper Limb Spasticity in Adults After Stroke or Traumatic Brain Injury. The study will be conducted in the U.S.A., approximately 128 adult subjects from approximately 30 study centers will be randomly assigned (1:1:1:1) to one of four treatment groups. The study consists of a 21-day screening period, a treatment visit and follow-up visits.

The protocol was amended and the study was completed with fewer subjects than described in the initial protocol due to impact of COVID-19 on enrollment.

DETAILED DESCRIPTION:
Subjects will be randomly assigned to DAXI for Injection 250 U, DAXI for Injection 375 U, DAXI for Injection 500 U, or placebo group, respectively. Eligible subjects will have ULS characterized by a primary aggregate posture

ELIGIBILITY:
Inclusion Criteria:

* 18 to 75 years of age
* Written informed consent including authorization to release health information
* Focal upper limb spasticity (ULS) after a stroke (as defined by WHO criteria) or traumatic brain injury (TBI), last stroke or TBI > 24 weeks prior to Screening
* ULS with the primary aggregate posture
* Moderate to severe ULS with a MAS score ≥ 2 at the elbow, wrist, and finger flexors
* Moderate to severe functional disability (Disability Assessment Score [DAS] score ≥2) on the principal target of treatment
* Has sufficient cognitive and communication ability to be able to give informed consent

Exclusion Criteria:

* Upper limb spasticity attributable to an etiology other than stroke or TBI.
* Bilateral upper limb paresis or quadriplegia.
* Initiated in physiotherapy of the upper extremities ≤ 30 days prior to Screening or planned to start physiotherapy of the upper extremities during the course of the study.
* Previous or planned treatment of the spastic upper limb with phenol, alcohol injection, or surgery
* Profound muscular atrophy or fixed contracture leading to marked limitation on range of motion
* Prior treatment with intrathecal baclofen
* Any neuromuscular neurologic conditions (amyotrophic lateral sclerosis, Lambert- Eaton, myasthenia gravis)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2018-12-12 (Actual); Primary Completion 2020-11-23 (Actual); Study Completion 2020-11-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (26):
- United States (26):
  - Rancho Research Institute at Rancho Los Amigos National Rehab Center, Downey, California
  - The Parkinsons and Movement Disorder Institute, Fountain Valley, California
  - Collaborative Neuroscience Network LLC, Long Beach, California
  - SC3 Research, Pasadena, California
  - Yale University, Fairfield, Connecticut
  - Waterbury Neurologists, Middlebury, Connecticut
  - Ki Health Partners LLC DBA New England Institute for Clinical Research, Stamford, Connecticut
  - MedStar National Rehabilitation Hospital, Washington D.C., District of Columbia
  - Parkinsons Disease and Movement Disorders Center, Boca Raton, Florida
  - NW FL Clinical Research Group, LLC, Gulf Breeze, Florida
  - Infinity Clinical Research, Hollywood, Florida
  - Parkinsons Disease Treatment Center of Southwest Florida, Port Charlotte, Florida
  - Shirley Ryan AbilityLab, Chicago, Illinois
  - Kansas Institute of Research, Overland Park, Kansas
  - William Beaumont Hospital, Royal Oak, Michigan
  - Rusk Rehabilitation Hospital, Columbia, Missouri
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Carolinas Rehabilitation, Charlotte, North Carolina
  - Wake Forest University School of Medicine, Salem, North Carolina
  - MossRehab, Elkins Park, Pennsylvania
  - University of Pittsburgh School of Medicine, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - North Texas Institute of Neurology and Headache, Frisco, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- DAXI 250 U: DAXI for injection for the treatment of Upper Limb Spasticity (ULS) in Adults with 250 U
Period: Overall Study
Arm/Group | DAXI 250 U | DAXI 375 U | DAXI 500 U | Placebo
Started | 22 | 19 | 18 | 24
Completed | 15 | 12 | 15 | 18
Not Completed | 7 | 7 | 3 | 6

BASELINE CHARACTERISTICS:
Population: Safety population
Groups:
- Total: Total of all reporting groups
Arm/Group | DAXI 250 U | DAXI 375 U | DAXI 500 U | Placebo | Total
Number analyzed (Participants) | 22 | 19 | 18 | 24 | 83
Age, Customized [Count of Participants; unit: Participants]
  <= 50 years | 10 | 6 | 5 | 7 | 28
  > 50 years | 12 | 13 | 13 | 17 | 55
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 10 | 5 | 12 | 34
  Male | 15 | 9 | 13 | 12 | 49
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 17 | 11 | 14 | 14 | 56
  Black | 4 | 6 | 3 | 10 | 23
  Asian | 1 | 1 | 0 | 0 | 2
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Other | 0 | 1 | 0 | 0 | 1
  Not provided | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline at Week 6 on the Modified Ashworth Scale (MAS) in the Suprahypertonic Muscle Group (SMG) Score
Description: Mean change from baseline at Week 6 in muscle tone measured with the Modified Ashworth Scale (MAS) in the Suprahypertonic Muscle Group (SMG) in one of the following: elbow, wrist, or finger flexors. Score range: 0 (Normal tone, no in tone) to 4 (Affected part{s} rigid in flexion or extension).
Time Frame: Week 6
Population: Intent to treat population
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | DAXI 250 U | DAXI 375 U | DAXI 500 U | Placebo
Number analyzed (Participants) | 22 | 19 | 18 | 24
score on a scale | -0.9 (0.25) | -1.0 (0.26) | -1.5 (0.27) | -0.8 (0.26)
Statistical Analysis 1: Comparison: DAXI 250 U vs Placebo; Test type: Superiority; p = 0.7645, ANCOVA
Statistical Analysis 2: Comparison: DAXI 375 U vs Placebo; Test type: Superiority; p = 0.5509, ANCOVA
Statistical Analysis 3: Comparison: DAXI 500 U vs Placebo; Test type: Superiority; p = 0.0488, ANCOVA

2. Primary Outcome: Physician Global Impression of Change (PGIC) Score
Description: Mean score on the Physician Global Impression of Change (PGIC) score at week 6. The PGIC is a single-item, 9-point scale that measures the physician's impression of improvement following treatment. Score range: -4 (Markedly worse) to +4 (Markedly improved).
Time Frame: Week 6
Population: Intent to treat population
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | DAXI 250 U | DAXI 375 U | DAXI 500 U | Placebo
Number analyzed (Participants) | 22 | 19 | 18 | 24
score on a scale | 1.5 (0.29) | 1.7 (0.30) | 1.7 (0.32) | 1.2 (0.28)
Statistical Analysis 1: Comparison: DAXI 250 U vs Placebo; Test type: Superiority; p = 0.3698, ANCOVA
Statistical Analysis 2: Comparison: DAXI 375 U vs Placebo; Test type: Superiority; p = 0.1972, ANCOVA
Statistical Analysis 3: Comparison: DAXI 500 U vs Placebo; Test type: Superiority; p = 0.2037, ANCOVA

3. Secondary Outcome: Muscle Tone Improvement Responder Rate
Description: Percentage of subjects who improve by a full point on the Modified Ashworth Scale (MAS) in the Suprahypertonic Muscle Group (SMG). Score range: 0 (Normal tone, no increase in tone) to 4 (Affected part(s) rigid in flexion or extension)
Time Frame: Weeks 6 and 12
Population: Intent to treat population
Measure: Count of Participants; unit: Participants
Arm/Group | DAXI 250 U | DAXI 375 U | DAXI 500 U | Placebo
Number analyzed (Participants) | 22 | 19 | 18 | 24
Participants
  Week 6 | 13 | 11 | 11 | 8
  Week 12 | 9 | 7 | 9 | 6

4. Secondary Outcome: Physician Global Impression of Change (PGIC) Responder Rate
Description: Percentage of subjects with improvement (i.e., a score of 1 to 4) on the Physician Global Impression of Change (PGIC). The PGIC is a single-item, 9-point scale that measures the physician's impression of improvement following treatment. Score range: -4 (Markedly worse) to +4 (Markedly improved). Scores of 1 or more indicate improvement following treatment.
Time Frame: Weeks 6 and 12
Population: Intent to treat population
Measure: Count of Participants; unit: Participants
Arm/Group | DAXI 250 U | DAXI 375 U | DAXI 500 U | Placebo
Number analyzed (Participants) | 22 | 19 | 18 | 24
Participants
  Week 6 | 17 | 16 | 14 | 15
  Week 12 | 15 | 17 | 13 | 13

5. Secondary Outcome: Change From Baseline at Weeks 6 and 12 on the Disability Assessment Scale (DAS) Functional Impairment
Description: Change from Baseline at Weeks 6 and 12 in functional impairment as measured by the Disability Assessment Scale (DAS) for the principal treatment target (PTT). DAS score range: 0 (No disability) to 3 (Severe disability - normal activities limited).
Time Frame: Weeks 6 and 12
Population: Intent to treat population
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | DAXI 250 U | DAXI 375 U | DAXI 500 U | Placebo
Number analyzed (Participants) | 22 | 19 | 18 | 24
score on a scale
  Week 6 | -0.9 (0.19) | -1.2 (0.19) | -0.7 (0.21) | -0.50 (0.20)
  Week 12 | -0.7 (0.21) | -1.0 (0.22) | -0.5 (0.21) | -0.8 (0.23)

6. Secondary Outcome: Duration of Effect
Description: Duration of effect is defined as time from injection (in weeks) until loss of muscle tone improvement in the SMG, as indicated by a reduction from baseline in MAS score of < 1-point and PGIC score is ≤ 0.
Time Frame: Up to 36 weeks
Population: Intent to treat population
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | DAXI 250 U | DAXI 375 U | DAXI 500 U | Placebo
Number analyzed (Participants) | 9 | 10 | 9 | 19
weeks | NA [13.0 to NA] — Insufficient subjects with an observed event | 24.0 [15.3 to NA] — Insufficient subjects with an observed event | 24.7 [5.7 to NA] — Insufficient subjects with an observed event | 8.4 [2.0 to 27.1]

7. Post Hoc Outcome: Change From Baseline at Week 4 in the Suprahypertonic Muscle Group (SMG) Score
Description: Mean change from baseline at Week 4 in muscle tone measured with the Modified Ashworth Scale (MAS) in the Suprahypertonic Muscle Group (SMG) in one of the following: elbow, wrist, or finger flexors. Score range: 0 (Normal tone, no in tone) to 4 (Affected part{s} rigid in flexion or extension).
Time Frame: Week 4
Population: Intent to treat population
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | DAXI 250 U | DAXI 375 U | DAXI 500 U | Placebo
Number analyzed (Participants) | 22 | 19 | 18 | 24
score on a scale | -0.9 (0.22) | -0.9 (0.23) | -1.8 (0.24) | -0.6 (0.22)
Statistical Analysis 1: Comparison: DAXI 250 U vs Placebo; Test type: Superiority; p = 0.4324, ANCOVA
Statistical Analysis 2: Comparison: DAXI 375 U vs Placebo; Test type: Superiority; p = 0.3893, ANCOVA
Statistical Analysis 3: Comparison: DAXI 500 U vs Placebo; Test type: Superiority; p = 0.0002, ANCOVA

8. Post Hoc Outcome: Change From Baseline at Week 4 in the Physician Global Impression of Change (PGIC) Score
Description: Change from Baseline at Week 4 in the Physician Global Impression of Change (PGIC). Score range: -4 (Markedly worse) to +4 (Markedly improved).
Time Frame: Week 4
Population: Intent to treat population
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | DAXI 250 U | DAXI 375 U | DAXI 500 U | Placebo
Number analyzed (Participants) | 22 | 19 | 18 | 24
score on a scale | 1.5 (0.24) | 1.7 (0.24) | 1.8 (0.26) | 0.9 (0.23)
Statistical Analysis 1: Comparison: DAXI 250 U vs Placebo; Test type: Superiority; p = 0.0562, ANCOVA
Statistical Analysis 2: Comparison: DAXI 375 U vs Placebo; Test type: Superiority; p = 0.0150, ANCOVA
Statistical Analysis 3: Comparison: DAXI 500 U vs Placebo; Test type: Superiority; p = 0.0092, ANCOVA

ADVERSE EVENTS:
Time Frame: The adverse events were collected throughout the entire study, up to 36 weeks.
Description: The Safety Population includes all subjects who received at least 1 study treatment injection and was used to assess AEs and SAEs
Arm/Group | DAXI 250 U | DAXI 375 U | DAXI 500 U | Placebo
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/19 | 0/18 | 0/24
Serious Adverse Events (participants affected / at risk) | 2/22 | 0/19 | 1/18 | 2/24
Other Adverse Events (participants affected / at risk) | 4/22 | 12/19 | 6/18 | 4/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DAXI 250 U (N=22) | DAXI 375 U (N=19) | DAXI 500 U (N=18) | Placebo (N=24)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coronavirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DAXI 250 U (N=22) | DAXI 375 U (N=19) | DAXI 500 U (N=18) | Placebo (N=24)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site bruising (General disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Injection site erythema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site hematoma (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site induration (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nail infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (3) | 0 (0) | 1 (1) | 0 (0)
Heat stroke (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urine analysis abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Myofascial pain syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cervical radiculopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nocturia (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study Center and/or Investigator shall submit to Revance a copy of the proposed publication at least sixty (60) days prior to the submission thereof for publication or disclosure to a third party: (i)to provide Revance with the opportunity to review and comment on the contents thereof, (ii)to identify any Confidential Information to be deleted from the proposed publication or disclosure, and (iii)or delay the publication or disclosure 90 days to allow Revance to pursue patent protections.

DOCUMENTS (2):
  • Study Protocol (2020-06-29): https://cdn.clinicaltrials.gov/large-docs/02/NCT03821402/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-11): https://cdn.clinicaltrials.gov/large-docs/02/NCT03821402/SAP_001.pdf